CLINICAL TRIAL: NCT06805149
Title: Evaluation of Emergency Computed Tomography in Suspected Renal Colic
Brief Title: Evaluation of Emergency Computed Tomography in Suspected Renal Colic. This is an Observational Retrospective Study Aimed to Evaluate Emergency Computed Tomography in Patients at the Emergency Department in Helsingborg, Sweden, With Suspected Acute Renal Colic.
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01345-01
Record Dates: First submitted 2025-01-15; First posted 2025-02-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-01

CONDITIONS: Kidney Stone
Keywords: Neprolithiasis; Kidney diseases; Urologic disease; Urinary calculi; Kidney calculi; Renal colic; Pain; Computed tomography; Urogenital disease
MeSH Terms: conditions — Kidney Calculi; Kidney Diseases; Urologic Diseases; Urinary Calculi; Renal Colic; Pain; Urogenital Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency CT: kidney stone?: Patients at the emergency department in Helsingborg with suspected acute renal colic with an CT within 24 hours.

SUMMARY:
The goal of this observational study is to learn more about diagnostics in patients with suspected acute renal colic at the emergency department. The main questions it aims to answer are:

* How many patients with symtoms of urolithiasis have a stone in the urinary tract at the emergency computed tomography (CT)
* Location and size of the stones.
* Evaluate time to intervention and closure and if this has changed due to emergency CT.

Participants are patients with symtoms of suspected acute renal colic at the emergency department in Helsingborg with an emergency CT within 24 hours.

DETAILED DESCRIPTION:
Since October 2022 The National Guidelines in Sweden recommend emergency CT for patients with suspected acute renal colic at the emergency department. In May 2023 the Department of Urology implemented this new regime with emergency CT for these patients in collaboration with the Department of Emergency and the Department of Radiology. This study aims to evaluate the first year (May 2023 to May 2024) with this new regime. Data regarding these patients where gathered regarding decriptive data, data regarding the stone, interventions and follow up. The investigators aim to compare the data with data from a soon to be published (Scandinavian Journal of Urology) article evaluating the situation regarding these patients during one year 2018-2019.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the emergency department with suspected acute renal colic and an emergency CT within 24 hours 10 May 2023 to 9 May 2024.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at the emergency department in Helsingborg
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Numbers of patients with a kidney stone on emergency CT | From enrollment until the date participants are considered stone free, up to 6 months regarding participants with stone. For participants without a stone, the time frame extends over the duration of their hospitalization, up to 30 days.
  Number of patients with a kidney stone on emergency CT. Size and location of the stone as well as time to intervention and closure for those with a stone.

SECONDARY OUTCOMES:
Numbers of visits to the emergency department | Time from enrollment until the date the participants are considered stone free, up to 6 months.
  Has the number of visits to the emergency department due to acute renal colic changed before and after implementation of emergencty CT

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Wagenius, Senior consultant, PhD, Principal Investigator — Urology Department Helsingborg
Locations (1):
- Urology Department, Helsingborg, Sweden

IPD SHARING:
Plan to Share IPD: No
We have no plans to share participants data outside the research group at the moment.